CLINICAL TRIAL: NCT05563285
Title: Effects of Exercise and Mindfulness-Based Intervention on Emotion Regulation and Inhibitory Control of Smartphone Addiction Among Female University Students
Brief Title: Effect of Exercise and MBI on Female Students' Emotion Regulation and Inhibitory Control of Smartphone Addiction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Huange Liu, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Huange Liu
Record Dates: First submitted 2022-09-25; First posted 2022-10-03 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Smartphone Addiction; Mental Health Issue
Keywords: Exercise; Mindfulness-Based Intervention; Smartphone Addiction; Emotion Regulation; Inhibitory Control; Female University Students
MeSH Terms: conditions — Internet Addiction Disorder; Motor Activity; Emotional Regulation | interventions — Exercise; Control Groups

STUDY DESIGN:
Intervention Model Description: In this experiment, the combination of Exercise and Mindfulness-Based Intervention method was used to intervene the smartphone addiction of female university students' emotion regulation and inhibitory control compared with the usual PE sessions method. Each parallel group has female separately.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise and Mindfulness-Based Intervention (Experimental): Patients in the intervention group will be provided exercise and mindfulness-based intervention was shown for the 1-8 weeks.
  Interventions: Behavioral: Exercise and Mindfulness-Based Intervention; Behavioral: Control Group
- Control Group (Active Comparator): Control group will not receive exercise and mindfulness-based intervention however, primary care service providers and mental health professionals will provide any required routine care according to their clinical judgment and available resources.
  Interventions: Behavioral: Exercise and Mindfulness-Based Intervention; Behavioral: Control Group

INTERVENTIONS:
Behavioral: Exercise and Mindfulness-Based Intervention — 1.Exercise Intervention
  1st-2nd week: 15 min for Brisk walking. Intensity: HRmax (60%-65%); CR10 (5-6). 3rd-4th week: 20 min for Brisk walking. Intensity:HRmax (65%-70%); CR10 (6-7). 5th-6th week: 25 min for Brisk walking. BW: Intensity: HRmax(70%-75%); CR10 (6-7). 7th -8th week:30 min for Brisk walking.
  Exercise Intervention basic content:
  (1) Gradually increase the walking speed; (2) Slowly reduce the speed; (3) Rest for 5 min.
  2. Mindfulness-Based Intervention
  1st-2nd week: 30 min for mindfulness training. 3rd-4th week: 35 min for mindfulness training. 5th-6th week: 40 min for mindfulness training. 7th-8th week: 45 min for mindfulness training.
  Mindfulness-Based Intervention basic content:
  (1) Yoga; (2) Mindful breathing; (3) Mindfulness meditation; (4) Body scan; (5) Mindfulness awareness; (6) RAIN technique; (7) Mindful Stretching; (8) Mindful walking; (9) Mindful running
Behavioral: Control Group — The control group maintained their classes as usual, usual physical education sessions, and usual daily life.

SUMMARY:
Mobile-based technology is advancing at an unprecedented rate, and in the past decade, smartphone use has become common among today's university students, who have mental health. A lot of attention has been paid in the media to the existence of "smartphone addiction" or problematic smartphone use(Sohn et al., 2019).Overuse of smartphones can cause health problems(Adams & Kisler, 2013; Demirci et al., 2015).

As an interdisciplinary subject, this study aimed at university students' smartphone addiction behavior research, understand the information era of college students' way of behavior patterns, exercise and psychological intervention strategy is put forward, to evaluate exercise and MBI intervention,and reduction of university students' smartphone addiction.

DETAILED DESCRIPTION:
This study was divided into two groups, the exercise and mindfulness-based intervention group, and the control group. This study evaluates the effect of 8-week exercise and MBI intervention on the capacity of emotional regulation measured by physiological and psychological state and inhibitory control of smartphone addiction in female university students. The sample was Chinese female university students aged 18-23 years with infrequent exercise for smartphone addiction.

According to the literature review, the frequency of brisk walking training in this experiment was scheduled for two times/week, with a total training duration of 8 weeks. Each training session was changed within two weeks. It ranged from 60 minutes in the first and second week to 90 minutes in the eighth week of the seventh week. Brisk walking was trained using maximum heart rate to control the intensity and measured using the Borg CR10 scale after training. All exercise techniques were taught before intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Female.
2. Aged 18 to 23.
3. Good health, no apparent speech disorder.
4. According to Leung's assessment scale, MAPI scores had to be more than 40 (out of 85) (Leung, 2008) .
5. .Without cardiovascular, metabolic, renal, or pulmonary diseases, symptoms, psychological disorders, or a history of alcohol abuse.And no participation in similar research projects before (using medication for psychiatric problems and undergoing other psychotherapeutic remedies)
6. Have time to ensure that you can attend every counseling on time.
7. They did no longer take part in any structured exercise in the past three months (e.g., walking, Tai Chi, basketball, badminton, running, yoga, weight training, etc.), and without experience of mindfulness training.
8. Subjects were able to participate and complete exercise training independently without any assistive devices.
9. Capable to be engaged, participate or respond to the research question,and willing to give informed consent.

Exclusion Criteria:

* Those who satisfy any of the following conditions shall be excluded:

  1. Mobile Phone Addiction Index (MPAI) scores below 40 They had major disease (respiratory illness, musculoskeletal disorder, dementia and metabolic, cardiovascular disease, and renal, or pulmonary diseases) and any psychosis or other severe psychiatric disorders. Records of extreme physical or psychological problems, which includes different addictive disorders, psychotic disorders, primary depression, borderline personality disorder, or antisocial character disease primarily based on the clinical psychologist's view or observations and oral questioning.
  2. Who are unable to move due to injury or illness and drop out of school .
  3. Those who were undergoing other psychotherapeutic treatments were also excluded from the study.
  4. Excluded students with sports contraindications and time conflicts.
  5. They have participated with exercise in the past three months (e.g., walking, running, weight training, etc.)

Ages: 18 Years to 23 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2022-12-25 (Estimated); Study Completion 2023-01-20 (Estimated)

PRIMARY OUTCOMES:
Mobile Phone Addiction Index (MPAI; Assessing Change) | Assessments will be conducted at baseline (after the screening), 4th week (1month) after the baseline, 8th week (2rd month)
  Smartphone addiction was assessed using the Mobile Phone Addiction Index (MPAI) (Leung, L. ,2008), which was translated into Chinese (Huang H,et,al.,2014) and is used widely in Chinese contexts (Zhao Y, 2019 & Chen Y,et,al.,2019). The MPAI contains 17 items assessing four domains: inability to control craving, feeling anxious and lost, withdrawal/escape, and productivity loss. Each item is responded to from 1 ("not at all") to 5 ("always"). Final scores were summed and higher total scores reflect higher levels of smartphone addiction. The Cronbach's alpha of the MPAI was 0.86 in the present study.
Smartphone behavior (Time spent on smartphone use; Assessing Change) | Assessments will be conducted at baseline (after the screening), 4th week (1month) after the baseline, 8th week (2rd month)
  Subjects (respondents) will answer through six relevant time categories. "Less than 10 minutes", "11-60 minutes", "1-2 hours", "3-4 hours", "5-6 hours", or "more than 6 hours". For the type of functionality of the smartphone software used, the subjects (respondents) used a 5-point Likert scale (0 = never, 1 = rarely, 2 = sometimes, 3 = usually, 4 = always).
Heart rate (HR; Assessing Change from physiological state) | Assessments will be conducted at baseline (after the screening), 4th week (1month) after the baseline, 8th week (2rd month)
  Heart rate is used to measure exercise intensity, and Emotion regulation involves emotional responses (physiological components) such as heart rate (HR).
Galvanic skin response (GSR; Assessing Change of physiological state) | Assessments will be conducted at baseline (after the screening), 4th week (1month) after the baseline, 8th week (2rd month)
  Emotion regulation involves emotional responses (physiological components) such as galvanic skin response (GSR)(Bosse, 2017).
Electroencephalography (EEG; Assessing Change of physiological state) | Assessments will be conducted at baseline (after the screening), 4th week (1month) after the baseline, 8th week (2rd month)
  Emotion regulation involves emotional responses (physiological components) such as electroencephalography (EEG).
Emotion Regulation Questionnaire (ERQ; Assessing Change) | Assessments will be conducted at baseline (after the screening), 4th week (1month) after the baseline, 8th week (2rd month)
  The Emotion Regulation Questionnaire (ERQ; Gross & John, 2003)
Positive and negative emotion scores (Assessing Change) | Assessments will be conducted at baseline (after the screening), 4th week (1month) after the baseline, 8th week (2rd month)
  Positive and negative emotion scores measured at different time points
Response Inhibition (Assessing Change of Inhibitory control) | Assessments will be conducted at baseline (after the screening), 4th week (1month) after the baseline, 8th week (2rd month)
  The measured variables were reaction time (RT) and accuracy.
Craving (Assessing Change) | Assessments will be conducted at baseline (after the screening), 4th week (1month) after the baseline, 8th week (2rd month)
  Craving for smartphones (modified desire for drinking questionnaire: Love, James,
  & Willner, 1998)

SECONDARY OUTCOMES:
Psychological Symptoms (Assessing Change) | Assessments will be conducted at baseline (after the screening), 4th week (1month) after the baseline, 8th week (2rd month)
  Psychological symptom using the Depression Anxiety Stress Scale-21 (DASS-21). to measure the emotional states (Oei et al., 2013) . This questionnaire is a short version of a self-report instrument (21 items) which measures depression, anxiety and tension/stress (negative emotional states).
Loneliness (Assessing Change) | Assessments will be conducted at baseline (after the screening), 4th week (1month) after the baseline, 8th week (2rd month)
  used the Chinese version of the ULS-8 loneliness scale, which was translated by Zhou et al. for participation in China.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Huange, Principal Investigator — University Putra Malaysia
Locations (1):
- Yulin University, Yulin, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No
Since this is my doctoral thesis experiment, I won't share it until I graduate.

REFERENCES:
- [Background] Billones R, Saligan L. What Works in Mindfulness Interventions for Medically Unexplained Symptoms? A Systematic Review. Asian Pac Isl Nurs J. 2020;5(1):1-11. doi: 10.31372/20200501.1082. PMID 32704524
- [Background] Chang YK, Labban JD, Gapin JI, Etnier JL. The effects of acute exercise on cognitive performance: a meta-analysis. Brain Res. 2012 May 9;1453:87-101. doi: 10.1016/j.brainres.2012.02.068. Epub 2012 Mar 4. PMID 22480735
- [Background] Fan H, Qi S, Huang G, Xu Z. Effect of Acute Aerobic Exercise on Inhibitory Control of College Students with Smartphone Addiction. Evid Based Complement Alternat Med. 2021 Aug 5;2021:5530126. doi: 10.1155/2021/5530126. eCollection 2021. PMID 34394381
- [Background] Garland EL, Howard MO. Mindfulness-based treatment of addiction: current state of the field and envisioning the next wave of research. Addict Sci Clin Pract. 2018 Apr 18;13(1):14. doi: 10.1186/s13722-018-0115-3. PMID 29669599
- [Background] Liu S, Xiao T, Yang L, Loprinzi PD. Exercise as an Alternative Approach for Treating Smartphone Addiction: A Systematic Review and Meta-Analysis of Random Controlled Trials. Int J Environ Res Public Health. 2019 Oct 15;16(20):3912. doi: 10.3390/ijerph16203912. PMID 31618879
- [Background] Stanton MV, Matsuura J, Fairchild JK, Lohnberg JA, Bayley PJ. Mindfulness as a Weight Loss Treatment for Veterans. Front Nutr. 2016 Aug 15;3:30. doi: 10.3389/fnut.2016.00030. eCollection 2016. PMID 27574603
- [Background] Zhou J, Wang L. Differences in the Effects of Reading and Aerobic Exercise Interventions on Inhibitory Control of College Students With Mobile Phone Addiction. Front Psychiatry. 2022 Mar 1;13:797780. doi: 10.3389/fpsyt.2022.797780. eCollection 2022. PMID 35299822